CLINICAL TRIAL: NCT05556954
Title: The Role of The Microbiome in Diabetic Foot Ulcers (DFU)
Brief Title: Diabetic Foot Ulcers Microbiome and Pathogen Identification
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brian Schmidt, Associate Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00214995; K23DK131261 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Foot Ulcer; Diabetes Mellitus; Wound
Keywords: Wound Infection; Wound assessments; Wound's microbiome
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus; Wounds and Injuries; Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infected DFU cohort: 25 participants that have an infected DFU will be enrolled.
  Interventions: Procedure: Wound debridement
- Non-infected DFU cohort: 75 non-infected participants with DFU will be enrolled.
  Interventions: Procedure: Wound debridement

INTERVENTIONS:
Procedure: Wound debridement — Participant that are having usual care visits for management of diabetic foot ulcers will be enrolled into this study. The procedure is done as part of standard of care. Tissue from the samples will be analyzed for this study.
  Aliquoting and Deoxyribonucleic acid (DNA) extraction will be done on the specimens. Bacterial DNA from biospecimens will be isolated, quantified, amplified, and sequenced.

SUMMARY:
This research is being done because people with diabetes have reduced healing capacity and prone to develop infections of foot wounds. This can be problematic because wounds that become infected may result in amputation and more severe complications. New evidence suggests that a better understanding of the microbiome of wounds (e.g., bacterial presence) may provide information about wound healing and provide an earlier opportunity to identify an individual who may be prone to develop diabetic foot infection in their wound.

Therefore, the purpose of this study is to evaluate the role of the microbiome of the diabetic foot ulcer in development of infection and wound healing. Once the role of the microbiome is confirmed, progress towards the prevention and treatment of diabetic foot ulcers and complications may be possible.

ELIGIBILITY:
Inclusion Criteria:

* DFU patients with diabetes mellitus
* Have a hemoglobin A1c[HbA1c] of 12% or less as measured within the last 6 months
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Pregnant or lactating
* Uncontrolled blood glucose as demonstrated by by a HbA1c of greater than 12%
* Bilateral wound or ulcer
* Current infection of Coronavirus (COVID-19)
* Unable to provide informed consent or are unwilling to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that are seen during usual care visits for management of diabetic foot ulcers in the University of Michigan (UM) Podiatry clinics within Metabolism, Endocrinology and Diabetes (MEND), the UM Comprehensive Wound Care Center, and from those consented participants in the Diabetic Foot Consortium (DFC) Biomarkers for Active Diabetic Foot Ulcers study,
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
The percent change in foot ulcer surface area (cm2) after 12 weeks of observation for either infected or non-infected diabetic foot ulcers | Baseline to 12 weeks

SECONDARY OUTCOMES:
The percent of clinically resolved infected DFU for infected diabetic foot ulcer participants | Baseline to 12 weeks
  Defined as improvement of greater or equal to 2 clinical signs (Local swelling or induration, erythema, local tenderness or pain, local warmth, purulent discharge) with no requirement for additional antibiotic(s).
Total days of antibiotic therapy for the DFU infected diabetic foot ulcer participants | Baseline to 12 weeks
Number of days to infection resolution for the DFU infected diabetic foot ulcer participants | Baseline to 12 weeks
The percentage of participants with an infected DFU at baseline that resolve clinical infection by study week 4 | Baseline to 4 weeks
Post-study percentage change of wound surface area (cm2) for both cohorts | Baseline to 12 weeks
Proportion of participants that reach a 50% reduction in surface area of the DFU for both cohorts | Baseline to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Schmidt, DPM, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No